CLINICAL TRIAL: NCT03910595
Title: An Efficacy Study of Mepitel Film in the Prophylaxis of Radiation-Induced Skin Reactions in Breast Cancer Patients Undergoing Adjuvant Radiotherapy
Brief Title: Efficacy Study of Mepitel Film the Prophylaxis of Radiation-Induced Skin Reactions in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Edward Chow, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 294-2018
Record Dates: First submitted 2019-01-24; First posted 2019-04-10 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer; Radiation Dermatitis
Keywords: Barrier Film; Mepitel; Quality of Life; Radiation Dermatitis; Skin toxicity
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis

STUDY DESIGN:
Intervention Model Description: All patients will receive the Mepitel film intervention. This film will be given to patients in one of three patient populations:
  1. Patients with large breasts
  2. Patients with small or medium sized breasts
  3. Patients with chest wall radiation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mepitel Film Arm (Experimental): This is a single arm trial where all patients will receive the intervention of Mepitel Film.
  Interventions: Other: Mepitel Film

INTERVENTIONS:
Other: Mepitel Film — Mepitel film is a barrier film that may help in reducing radiation dermatitis by limiting friction.

SUMMARY:
In patients undergoing adjuvant radiotherapy for breast cancer, radiation-induced skin toxicities are a common occurrence and adversely impact patients' quality of life (QOL). In the last decade, there have been no significant advances in preventing or treating radiation-induced skin toxicities. Recently, a phase III randomized trial by Herst et al. (n=78) in New Zealand showed that the prophylactic use of Mepitel Film reduced skin reaction severity by 92% compared to skin treated only with aqueous cream. Mepitel film has not been widely adopted in North America. To validate the efficacy of the film and guide the development of a larger multi-centre phase II study, a pilot study testing the efficacy of the film is proposed. In the study, 30 patients will have the film applied on their breast for the duration of radiation treatment and their skin reactions will be assessed throughout the treatment and after the treatment. The investigators hypothesize that the severity and incidence rates of skin reactions for patients using Mepitel film will be lower when compared to real world data from our centre, and that cosmetic outcomes will be improved with the film.

DETAILED DESCRIPTION:
In patients undergoing adjuvant radiotherapy for breast cancer, radiation-induced skin toxicities are a common occurrence and adversely impact patients' quality of life (QOL). Patients with large breasts or patients receiving chest wall radiation may be more likely to have worse skin reactions following radiation. In the last decade, there have been no significant advances in preventing or treating radiation-induced skin toxicities. Recently, a phase III randomized trial by Herst et al. (n=78) in New Zealand showed that the prophylactic use of Mepitel Film prevented moist desquamation (26% vs. 0%, p < 0.001) and reduced skin reaction severity by 92% (p < 0.001) compared to skin treated only with aqueous cream. Another study by Moller et al. (n=101) in Denmark reported a non-significant improvement in observer-rated radiation dermatitis with the film (p=0.1) compared to cream, and significant improvements in several patient-reported outcomes. Moreover, patients with breast cancer complain of hyperpigmentation in the radiated area during and after radiation.

Mepitel Film has not been widely adopted in North American clinical practice. To further study and validate the efficacy of Mepitel Film in preventing acute skin reactions caused by breast radiation and elucidate its efficacy in preventing poor cosmetic outcomes, a phase II efficacy study of three patient populations will be conducted:

1. Patients with large breasts
2. Patients with small or medium sized breasts
3. Patients with chest wall radiation

The results of the phase II efficacy study can guide the development of a subsequent multi-centre phase II and III trials to further validate the use of Mepitel film and increase its adoption rate.

The primary objective is to examine the efficacy of Mepitel film in the prophylaxis of radiation-induced skin reactions. Secondary objectives include an evaluation of patient-reported and healthcare professional (HCP)-reported skin toxicities including moist desquamation with the use of Mepitel film.

Radiation oncologists will first introduce the study to their patients in their breast clinic, showing a sample of the product and also pictures from the trial conducted in New Zealand. Patients if interested may be provided a patient information sheet to review at home. Then, patients will be approached by a CRA at their radiation planning appointment to review all information and obtain informed consent.

All patients will receive Mepitel film for the duration of treatment. Radiation treatment will be delivered as prescribed by the treating radiation oncologist and may include a variety of techniques and beam modifiers.

Trained clinical research assistants (CRA) or the radiation review nurse will apply the Mepitel film for patients prior to their first radiation treatment at a designated clinic room and will check daily prior to radiation that the breast/chest wall has not been distorted by the film. If the film needs to be readjusted, the CRAs or nurses will remove peeling sections of film and reapply where needed. The film will be removed two weeks post radiation treatment.

Patients will complete evaluations once a week at their regular review clinic visit and will be assessed by an HCP or CRA. At the last treatment or last review appointment, a photo of the patient's breasts/chest wall will be taken, and they will be asked to complete an assessment. An HCP will also conduct an assessment.

After completion of radiation, patients will be called at week 1 and weeks 3-6 to assess endpoints. Patients will be asked to return for a 2-week, 3-month, and 6-month follow-up assessment where photos of their breasts/chest wall will be taken, and they will complete their personal assessments. The film will be removed at the 2-week follow-up appointment. The 3-month follow-up assessment will occur at the same time as their regular clinic follow-up with their radiation oncologist. At the 3-month and 6-month follow-up assessment, an HCP will also an assessment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Patient will receive adjuvant breast or chest wall radiation
* Post-lumpectomy patients with band size of at least 36 inches or cup size of D or larger will be part of the large breast cohort
* Post-lumpectomy patients that do not meet this size requirement will be part of the small or medium sized breast cohort
* Post-mastectomy patients are part of the chest wall radiation cohort
* Can communicate in English or be aided by a hospital translator

Exclusion Criteria:

* Patient had previous radiation therapy to the treatment area
* Patient had breast reconstruction
* Patient has a Karnofsky Performance Status score <70
* Patient will have radiation treatment in prone or reverse decubitus positions
* Patient will receive partial breast external beam radiation or brachytherapy
* Patient will receive radiation to the supraclavicular region

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-09-08 (Actual)

PRIMARY OUTCOMES:
Observable differences between treated and non-treated breasts/chest wall | Within 3 months following radiation
  Determined by a cosmetic dermatologist from photographs of the treated and non-treated breast/chest wall.

SECONDARY OUTCOMES:
Patient reports of acute skin toxicity | Within 3 months following radiotherapy
  Measured by the Skin Symptom Assessment (SSA); subscales for itchiness, pain/soreness, blistering/peeling, redness, discolouration/darkness, swelling, and trouble fitting brassieres graded as "not at all", "a little", "quite a bit", or "very much"
Patient reports of late skin toxicity | 6 months following radiotherapy
  Measured by the SSA; subscales for itchiness, pain/soreness, blistering/peeling, redness, discolouration/darkness, swelling, and trouble fitting brassieres graded as "not at all", "a little", "quite a bit", or "very much"
Clinician reports of acute skin toxicity | Within 3 months following radiotherapy
  Measured by the SSA; subscales for itchiness, pain/soreness, blistering/peeling, redness, discolouration/darkness, swelling, and trouble fitting brassieres graded as "not at all", "a little", "quite a bit", or "very much"
Clinician reports of late skin toxicity | 6 months following radiotherapy
  Measured by the SSA; subscales for itchiness, pain/soreness, blistering/peeling, redness, discolouration/darkness, swelling, and trouble fitting brassieres graded as "not at all", "a little", "quite a bit", or "very much"
Clinician grading of acute skin toxicity | Within 3 months following radiotherapy
  Measured by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE); graded on a scale from 0 (best) to 4 (worst)
Clinician grading of late skin toxicity | 6 months following radiotherapy
  Measured by the NCI CTCAE; graded on a scale from 0 (best) to 4 (worst)
Degree of acute skin toxicity and interference with daily functioning | Within 3 months following radiotherapy
  Measured by the Radiation Induced Skin Reaction Assessment System (RISRAS); researcher subscales for erythema and dry desquamation rated from 0 (best) to 4 (worst); researcher subscale for moist desquamation rated from 0 (best) to 6 (worst); researcher subscale for necrosis rated from 0 (best) to 10 (worst); patient subscales for tenderness/discomfort/pain, itchiness, burning sensation, and interference with daily activities rated from 0 (best) to 3 (worst).
Degree of late skin toxicity and interference with daily functioning | 6 months following radiotherapy
  Measured by the RISRAS; researcher subscales for erythema and dry desquamation rated from 0 (best) to 4 (worst); researcher subscale for moist desquamation rated from 0 (best) to 6 (worst); researcher subscale for necrosis rated from 0 (best) to 10 (worst); patient subscales for tenderness/discomfort/pain, itchiness, burning sensation, and interference with daily activities rated from 0 (best) to 3 (worst).
Long-term changes in skin pigmentation | Changes from baseline to 6 months following radiotherapy
  Measured by photographs of the treated and non-treated breast and graded by a cosmetic dermatologist
Acute changes in breast cosmesis | Within 3 months following radiotherapy
  Measured by the European Organization for Research and Treatment of Cancer (EORTC) Breast Cosmetic Rating System; subscales for breast size, breast shape, location of areola/nipple, shape of areola/nipple, tanning, pallor, breast edema, appearance of scar, and telangiectasia graded from 0 (best) to 3 (worst); overall grade assigned from 0 (best) to 2 (worst).
Late changes in breast cosmesis | 6 months following radiotherapy
  Measured by the EORTC Breast Cosmetic Rating System; subscales for breast size, breast shape, location of areola/nipple, shape of areola/nipple, tanning, pallor, breast edema, appearance of scar, and telangiectasia graded from 0 (best) to 3 (worst); overall grade assigned from 0 (best) to 2 (worst).
Film Integrity Assessment | Until film is removed, 2 weeks following radiotherapy
  Evaluated daily prior to the patient's radiotherapy treatment

CONTACTS AND LOCATIONS:
Overall Officials: Edward LW Chow, MBBS, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada